CLINICAL TRIAL: NCT01509209
Title: Efficacy and Safety of Cossac L Tablet in Vasomotor Rhinitis Patients : A Randomized, Double-blind, Placebo-controlled, Phase 3 Clinical Trial
Brief Title: Efficacy/Safety of Pseudoephedrine Plus Levocetirizine Versus Placebo in Patients With Vasomotor Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-LCT-301
Record Dates: First submitted 2012-01-10; First posted 2012-01-12 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Vasomotor Rhinitis
Keywords: vasomotor; pseudoephedrine; levocetirizine
MeSH Terms: conditions — Rhinitis, Vasomotor | interventions — Pseudoephedrine; levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Pseudoephedrine / Levocetirizine
- Cossac L (Experimental): Pseudoephedrine 120mg + Levocetirizine 2.5mg
  Interventions: Drug: Pseudoephedrine / Levocetirizine

INTERVENTIONS:
Drug: Pseudoephedrine / Levocetirizine — tablet, BID everyday
  Other Names: Cossac L

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Cossac L tablet in the treatment of vasomotor rhinitis

DETAILED DESCRIPTION:
randomized, double-blind, placebo-controlled, phase 3

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of vasomotor rhinitis

Exclusion Criteria:

* Significant concomitant medical condition
* Use corticosteroids or other allergy medications during the study
* Considered by investigator as not appropriate to participate in the clinical study with othe reason

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
TVRSS(Total Vasomotor Rhinitis Symptom Score) | 2week
  the change from baseline in TVRSS

SECONDARY OUTCOMES:
TVRSS, VRSS | 1week or 2 week
  * the change from baseline in TVRSS during 1st week and 2nd week
  * the change from baseline in each vasomotor rhinitis symptom score at overall, during 1st week/2week

CONTACTS AND LOCATIONS:
Overall Officials: Kyungmi Park, Ph.D., Study Director — Hanmi Pharmaceutical Company Limited
Locations (1):
- ear, nose and throat, Boramae Hospital, Dongjak, Seoul, South Korea